CLINICAL TRIAL: NCT00924599
Title: Prevention of Gestational Diabetes Pilot Study
Brief Title: A Pilot Study Using Weightloss and Exercise to Prevent Recurring Gestational Diabetes in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Associate Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP-GDPP
Record Dates: First submitted 2009-05-04; First posted 2009-06-19 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Gestational Diabetes
Keywords: Recurring Gestational Diabetes; Prevention
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention Group-English (Experimental): Intervention Group will be learning how to lose weight through healthy eating and moderate exercise. The goal is to get participants to lose 7% of body weight and increase physical activity to 2 1/2 hours per week. This group will be meeting one time per week for twelve weeks, and then one time per month until conception.
  Interventions: Behavioral: Prevention of recurrent gestational diabetes through weight loss and exercise (English & Spanish)
- Intervention Group-Spanish (Experimental): Intervention Group will be learning how to lose weight through healthy eating and moderate exercise. The goal is to get participants to lose 7% of body weight and increase physical activity to 2 1/2 hours per week. This group will be meeting one time per week for twelve weeks, and then one time per month until conception.
  Interventions: Behavioral: Prevention of recurrent gestational diabetes through weight loss and exercise (English & Spanish)
- Lifestyle education-English (Active Comparator): The lifestyle education group will focus on learning about healthy eating, and healthy activity. This group will also learn stress reduction techniques as well as new ways of increasing activity. Group will meet one time per month for 3 months, then once a month until conception.
  Interventions: Behavioral: Lifestyle education (English & Spanish)
- Lifestyle education-Spanish (Active Comparator): The lifestyle education group will focus on learning about healthy eating, and healthy activity. This group will also learn stress reduction techniques as well as new ways of increasing activity. Group will meet one time per month for 3 months, then once a month until conception.
  Interventions: Behavioral: Lifestyle education (English & Spanish)

INTERVENTIONS:
Behavioral: Prevention of recurrent gestational diabetes through weight loss and exercise (English & Spanish) — Intervention groups will attend weekly sessions focused on healthy weight loss, healthy eating, exercise.
  Arms: Intervention Group-English; Intervention Group-Spanish
Behavioral: Lifestyle education (English & Spanish) — The lifestyle education group will focus on learning about healthy eating, and healthy activity. This group will also learn stress reduction techniques as well as new ways of increasing activity. Group will meet one time per month for 3 months, then once a month until conception.
  Arms: Lifestyle education-English; Lifestyle education-Spanish

SUMMARY:
The purpose of this study is to examine the feasibility of recruiting and providing a behavioral weight loss program prior to pregnancy to reduce gestational diabetes recurrence.

ELIGIBILITY:
Inclusion Criteria:

* GDM in last pregnancy
* BMI 30-40
* Age 18-40
* 1-5 years since last pregnancy
* Non-smoking
* English or Spanish speaking
* Planning to have a baby but willing to use birth control during the 3 month weight loss program

Exclusion Criteria:

* 3 or more miscarriages
* History of infertility
* Type 1 or Type 2 diabetes
* Any weight loss since last pregnancy (based on last pre-pregnancy weight)
* History of major psychiatric illness, drug abuse, or unsafe dieting practices
* History of bariatric surgery, major medical conditions that prohibit physical activity or dietary intervention (MD consent may be required)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes not present in pregnancy | from conception to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD., Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- Sierra Vista Regional Medical Center, San Luis Obispo, California, United States